CLINICAL TRIAL: NCT00760682
Title: Hyperbaric Oxygen Treatment of Mandibular Osteoradionecrosis. A Randomized Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lone Forner (Other)
Responsible Party: Sponsor-Investigator, Lone Forner, DDS, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 21
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Osteoradionecrosis
Keywords: osteoradionecrosis; hyperbaric oxygen; sequestrectomy
MeSH Terms: conditions — Osteoradionecrosis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 30 preoperative HBO sessions, sequestrectomy and 10 postoperative HBO sessions. The duration of each session is 90 minutes. 100 % oxygen is inhaled during decompression to 2.4 ATA.
  Interventions: Procedure: Hyperbaric oxygen
- 2 (No Intervention): Sequestrectomy without HBO treatment

INTERVENTIONS:
Procedure: Hyperbaric oxygen — 30 preoperative and 10 postoperative HBO sessions 90 minutes each. Sequestrectomy is performed after 30 sessions.
  Arms: 1

SUMMARY:
There is currently not sufficient evidence that hyperbaric oxygen (HBO) benefits the surgical removal of necrotic bone in osteoradionecrosis patients. This study aims at testing the hypothesis that HBO does improve healing after surgical removal of necrotic bone in irradiated previous head and neck cancer patients compared to not receiving HBO.

DETAILED DESCRIPTION:
1. Study objective

   The objective of the study is to evaluate the effect of hyperbaric oxygen (HBO) on mandibular osteoradionecrosis as an adjunctive to surgical treatment in patients previously irradiated for head and neck cancer.

   Hypothesis: Osteoradionecrosis lesions heal more frequently when administering HBO as an adjunct to surgery.
2. Introduction and rationale

   Each year, 300 danish patients are diagnosed with oral cancer. The majority of these cancers are planocellular carcinomas. The established treatments are surgery and radiation therapy. Depending on multiple factors such as total radiation dose, fractionation, localization and use of brachytherapy, mandibular osteradionecrosis occurs in 5-15% of previously head and neck irradiated patients.

   Osteradionecrosis is defined by National Cancer Institute (NCI) as radiation-induced cell death in components of bone (e.g., the marrow fat and mineralized tissue). It represents the final common pathway of several disease entities, which result in impaired blood supply to the bone tissue causing bone necrosis. Often, osteoradionecrosis is clinically expressed in relation to surgery or a similar tissue trauma, but may also arise spontaneously several years after radiation treatment. Oral rehabilitation is difficult in these patients as denture wear is painful. Furthermore, radiation-induced hyposalivation complicates retention of dentures, which are normally retained by a thin saliva film. As denture wear appears difficult, insertion of implants seems obvious in these patients. However, the survival rate of dental implants are reduced when inserted in irradiated bone. Thus, osteoradionecrosis patients has great requirements regarding pain therapy as well as oral functional and social rehabilitation.

   HBO is currently offered to osteoradionecrosis patients as a standard treatment in combination with surgical removal of the necrotic bone (sequestrectomy). 30 preoperative and 10 postoperative treatment sessions are given daily (on weekdays) during eight weeks. The duration of each treatment session is 90 minutes and involves inhalation of 100% oxygen during decompression to 15 meters (2.5 ATA). The decompression leads to an increased oxygen tension in the tissues. HBO stimulates monocyte and fibroblast proliferation as well as collagen synthesis in irradiated tissue. Also, angiogenesis is stimulated, resulting in an increased vascularity. Moreover, recent research shows that HBO induces bone marrow derived progenitor cells in previously irradiated humans and animals.

   At this point, there is not sufficient scientific evidence for a clinical effect of HBO on osteoradionecrosis. The majority of relevant studies are casuistic reports and case-control studies with few participants. Few randomized clinical trials (RCT) have been conducted. Two of these studies document an effect of HBO, but one of the studies only include twelve participants, which is not associated with sufficient power. The other study document a prophylactic effect of HBO on osteoradionecrosis, and does therefore not conclude on any treatment effects. The authors of the third study conclude, that there is no effect of HBO treatment. However, in this study, the protocol was closed before full inclusion (68 vs. 222), and therefore, the power may not be sufficient. Furthermore, the study protocol lacks accordance with the standard HBO protocol and sufficient description of the surgical interventions. Moreover, there is an unrealistically high recovery rate in the control group with following risk of drawing the wrong conclusions.

   A Cochrane review states that there is not sufficient amounts of data to perform a meta-analysis. Thus, more randomized clinical studies are needed in order to document whether there is an effect of HBO on osteoradionecrosis.
3. Endpoints

   3.1. Primary endpoint The primary endpoint recovery from osteoradionecrosis as defined by the NCI Common Toxicity Criteria of Adverse Events (CTCAE) v 3.0. Recovery is defined as no signs of osteoradionecrosis according to these criteria or grade 1 on this scale.

   Grade 1: Asymptomatic, radiographic findings only. Grade 2: Symptomatic and interfering with function, but not interfering with ADL (Activities of Daily Living , , , ). Minimal bone removal indicated i.e. minor sequestrectomy)..

   Grade 3: Symptomatic, interfering with ADL. Operative intervention or hyperbaric oxygen indicated.

   Grade 4: Disabling Grade 5: Death

   3.2. Secondary endpoints
   * Life quality (EORTC schemes QLQ-C30, QLQ-H&N35)
   * Body Mass Index
   * Pain intensity (VAS)
   * Analgetics consumption
   * Antibiotics consumption
   * Trismus
   * Xerostomia
   * Dysphagia
   * Dental status

   CTCAE v. 3.0 is based on clinical as well as ADL related criteria. The primary endpoint value is obtained by filling out 21-05 and 21-06. The ORN stadium is the highest obtained score. In patients not wearing dentures, the denture-related question can be omitted.
4. Investigational plan

   4.1. Inclusion

   All patients eligible for the study will be asked for informed consent by the protocol responsible person. If the patient does not wish to participate in the study, standard treatment will be given (HBO and surgery). Verbal and written information about the study will be given during the preliminary investigation. Randomization will occur approximately one week prior to participation.

   4.1. Study plan

   After confirmation of study eligibility, the participant is randomized to either group I (HBO and surgery) or group II (surgery).

   Drug registration is performed at home until 3 months postsurgically. After this point, information is obtained from a central register.

   The study is not blinded, as we consider it unrealistic to blind the investigator because of risk of 1) the participant unintentionally mentions details from the HBO treatment or that the investigator runs into the patient at the hyperbaric facility.

   The trials is ended when 114 participants are included. Participants withdrawn from the study will be replaced until 114 have completed participation. A drop-out rate of 20-30% is considered likely, which means that in total, 150 potential participants will be asked to participate in order to obtain 114 observations. The drop-out The drop-out rate will be evaluated throughout the study. All patients eligible for the study will be asked for informed consent by the protocol responsible person. If the patient does not wish to participate in the study, standard treatment will be given (HBO and surgery). Verbal and written information about the study will be given during the preliminary investigation. Randomization will occur approximately one week prior to participation.
5. Prior to participation

Prior to inclusion, the participants is examined by a hyperbaric physician and a head and neck surgeon to ensure that the following criteria are met.

Inclusion criteria

1. Osteoradionecrosis grade 2, 3 or 4 (CTCAE v 3.0.)
2. Localization: Mandibula
3. Age > 18 No contraindications for hyperbaric oxygen treatment, e.g. emphysema, uncontrolled asthma, epilepsy, previous optic neuritis

Exclusion criteria solely applies for HBO treatment. Should any criteria arise after the HBO treatment, it is unnecessary to withdraw the patient from participation.

1. Malignancy/residual cancer
2. Previous HBO treatment
3. Pregnancy or lactation (fertile female participants are required to use safe anticonception)
4. Unmanageable claustrophobia
5. Undrained pneumothorax
6. Uncontrollable hypertension or blood pressure >220/110
7. Explosion of titanium reconstruction device

   5.2. Clinical evaluation prior to treatment

   Examination at baseline is carried out using the existing HBO examination programme and includes following anamnestic registrations:

   § Epilepsy

   § Lung disease

   § Heart disease

   § Diabetes
   * Psychologic or psychiatric disorders (to evaluate the need for medication during HBO)
   * Drug list
   * Use of eyeglasses

   Objective examination

   § Ability to equalize the pressure in the ears and sinuses (otherwise drained)

   § Heart and lung stetoscopy
   * Blood pressure
   * Weight
   * Pain assessment (VAS)

   5.3. Inclusion, randomization and stratification. For all eligible patients with informed consent, a DAHANCA 21-inclusion form, which is a checklist for inclusion- and exclusion criteria is filled out and faxed to the DAHANCA office: Fax +45 86 19 71 09. The fax is returned with randomization number and treatment regimen.

   Included patients will be stratified according to
   * Gender
   * ORN stadium

6. Treatment

All patients will be followed closely during their treatment. The investigator will perform the evaluations blinded. Since HBO treatment is time-consuming (8 weeks) and expensive (2000 DKK per session), it is not possible, nor ethically acceptable, to include a placebo group in order to conduct the study blinded to the participants.

6.1. Hyperbaric oxygen treatment

The patient will be decompressed according to a standard profile used in the clinic. During the first five minutes, the patient is decompressed to 14,5 +/- 0,5 m (2,45 +/- 0,05 ATA) and stays here for the next 90 minutes. Decompression to the surface (0 m) will hereafter take place during five minutes. The patient will breathe 100% oxygen during the full 100-minute procedure inside a hood (Amron Systems, California, USA) or mask (Divex Hyperlite II (Divex Industries, Aberdeen, Scotland). Each patient receives 30 preoperative treatment and 10 postoperative treatments.

6.2. Surgical treatment

All patients with ORN grade >1 will be surgically treated according to standardized guidelines. The interventions implies either

1. Resection of necrotic bone (sequestrectomy) with preservation of mandibular continuity.
2. Resection of necrotic bone (sequestrectomy) with loss of mandibular continuity. The least mutilating intervention will be performed. Resection with loss of continuity will only be performed in case of potential or stated fracture.

6.3. Termination of participation

Protocol treatment will be terminated in case:

The patient wish to terminate participation. New indication for surgery arises because of osteoradionecrosis at another localization.

Other unintentional events occurs that may impede participation.

7. Clinical evaluation and follow-up

7.1. One week after sequestrectomy The first evaluation occurs one week after surgery in order to evaluate wound healing.

7.2. One month after sequestrectomy (+/- two weeks).

7.3. Three months after sequestrectomy (+/- three weeks).

7.4. One year after sequestrectomy (+/- one month).

7.5. After relapse/progression In case of relapse or progression patients are treated according to local guidelines.

7.6 Follow-up

All patients are followed once a year for at least 5 years after completion of participation. Additionally, patients are instructed to contact the department in case of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Osteoradionecrosis grade 2, 3 or 4 according to the CTCAE v 3.0 criteria
* Localized to the mandibula
* > 18 yrs old

Exclusion Criteria:

* Existing malignant disease
* Previous HBO
* Pregnancy or lactation
* Uncontrollable claustrophobia
* Undrained pneumothorax
* Blood pressure > 220/110
* Exposed titanium reconstruction device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2008-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Osteoradionecrosis status according to the National Cancer Institute Common Toxicity Criteria v 3.0 | 1 year

SECONDARY OUTCOMES:
Life Quality | 1 year
  EORTC QoL-30 and H&N35
Body mass index | 1 year
  Body mass index
Pain intensity | 1 year
  Pain intensity on a VAS scale and based on analgetics consumption
Trismus | 1 year
  Ability to open the mouth
Xerostomia | 1 year
  Questionnaire
Dysphagia | 1 year
  Dysphagia according to the National Cancer Institute Common Toxicity Criteria v 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Lone Forner, DDS, PhD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (4):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Department of Anaesthesia, Copenhagen University Hospital, Copenhagen
- Sahlgrenska Universitet, Gothenburg, Sweden
- Aintree University Hospital, Liverpool, United Kingdom

REFERENCES:
- See also: Related Info — http://www.hbo.dk